CLINICAL TRIAL: NCT07182981
Title: Investigating the Relationship Between the Biopsychosocial Status of Patients Diagnosed With Scleroderma and Their Chewing and Swallowing Performance
Brief Title: Patients Diagnosed With Scleroderma and Their Chewing and Swallowing Performance
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 25/528
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Systemic Sclerosis (SSc); Scleroderma; Scleroderma (Limited and Diffuse); Scleroderma, Localized; Swallowing
Keywords: Juvenile scleroderma; scleroderma; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Localized; Juvenile-onset scleroderma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases diagnosed with scleroderma: Child and adult scleroderma patients who visited the rheumatology outpatient clinic at a university hospital will complete a questionnaire.
  Interventions: Other: Questionnaire application for child and adult scleroderma patients

INTERVENTIONS:
Other: Questionnaire application for child and adult scleroderma patients — Scales will be applied to cases diagnosed with scleroderma

SUMMARY:
It is recommended to focus on the physical functionality, chewing, and swallowing performance of individuals diagnosed with scleroderma. There is a need to address children and adults diagnosed with scleroderma comprehensively and to evaluate them on a biopsychosocial basis to support their disease management. The aim was to assess the biopsychosocial characteristics of both children and adults diagnosed with scleroderma and to examine their chewing and swallowing performance.

Additionally, this study aims to identify effective scales that can be used in future research to assess chewing and swallowing in individuals diagnosed with scleroderma.

ELIGIBILITY:
For a child diagnosed with scleroderma:

Inclusion Criteria:

* Cases diagnosed with scleroderma,
* Cases aged 7-18 years will be included.

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease, and malignancies
* Cases that are not willing to participate in the study will be excluded.
* Having participated in a regular exercise program for the past 3 months
* Individuals who are not willing to participate in the study

For adults diagnosed with scleroderma:

Inclusion Criteria:

* Individuals diagnosed with scleroderma,
* Individuals over the age of 18 will be included.

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease, and malignancies
* Individuals who are not willing to participate in the study will be excluded.
* Having participated in a regular exercise program for the past 3 months
* Individuals who are not willing to participate in the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
Pediatric Eating Assessment Scale (PEDI-EAT-10) | Two weeks
  It is used to evaluate swallowing disorders in pediatric patients. It was developed as the pediatric version of the EAT-10, which is used in adults. The PEDI-EAT-10 comprises 10 questions, each with a Likert scale ranging from 0 to 4 (0 = no problem, 4 = severe problem). The total score is calculated out of 40 points.
Chewing and Swallowing Test for Children (TOMASS-C) | Two weeks
  It is a measurement tool developed specifically for children to assess chewing performance. TOMASS-C is a standardized method that quantitatively evaluates the chewing and swallowing of a solid food (cracker) in the pediatric population. During the test, the following parameters will be observed and recorded:
  * Number of bites
  * Number of chewing cycles
  * Number of swallows
  * Task completion time (in seconds)
3-Ounce Water Swallow Challenge | Two weeks
  It is a commonly used method for assessing oropharyngeal dysphagia and aspiration risk. Subjects must swallow 3 ounces (90 cc) of water without interruption. Failure to complete the task, coughing, choking, or exhibiting a wet-gurgling voice quality within 1 minute during or after the test is included. Subjects who can drink 90 cc of water completely and in one go without coughing, choking, or drinking the water in portions have completed the test.
Turkish Eating Assessment Tool (T-EAT-10) | Two weeks
  It is a questionnaire consisting of 10 questions with a Likert scale ranging from 0 to 4 (0 = no problem, 4 = severe problem). The total score is calculated out of 40 points by summing the responses given to each question. A score of 3 or higher is considered abnormal in the questionnaire.
Test of Masticating and Swallowing Solids (TOMASS) | Two weeks
  The test evaluates how many bites it takes an individual to eat a biscuit while sitting upright, how many chewing cycles they perform, how many times they swallow, and the total time from bite to swallow. The number of bites, number of chewing cycles, number of swallows, and total time will be calculated.
Maximum Mouth Opening (MMO) | Two weeks
  After ensuring that individuals open their mouths as wide as possible, the distance between the incisal edges of the central incisors in the upper and lower jaws will be measured in millimeters using a ruler, and the values will be recorded.
Dysphagia Limit (DL) | Two weeks
  Individuals are given liquids in volumes of 5, 10, 15, 20, 25, 30, 35, 40, and 45 mL using a graduated syringe, and they are asked to swallow the liquid. The maximum amount of liquid that can be swallowed during a single movement of the thyroid cartilage is determined. In healthy individuals, the normal dysphagia limit is more than 20 mL. If a person can normally swallow 20 mL, the dysphagia limit is considered normal.

SECONDARY OUTCOMES:
Modified Rodnan skin score (MRSS) | Two weeks
  A pediatric and adult rheumatologist assessed it. The MRSS evaluates skin thickening in 17 body regions, graded from 0 (normal) to 3 (severe skin thickening). The total score ranges from 0 to 51, with increased scores indicating poor skin involvement.
Localized Scleroderma Assessment Tool (LoSCAT) | Two weeks
  LoSCAT consists of two sections: the modified Localized Skin Severity Index, which measures disease activity, and the Localized Scleroderma Damage Index, which assesses damage (usually scored between 0 and 3). In the Localized Skin Severity Index, it evaluates the color of the lesion border for erythema, skin thickness, and the presence of new lesions or lesion extension. In the Localized Scleroderma Damage Index, three areas of cutaneous damage are combined to obtain a score. These areas evaluate hyperpigmentation or hypopigmentation, whichever is more prominent, as well as dermal atrophy, subcutaneous atrophy, and dyspigmentation.
Mouth Handicap in Systemic Sclerosis Questionnaire (MHIIS) | Two weeks
  It consists of 12 items. Each item is scored from 0 to 4, with response options of "Never (0)", "Rarely (1)", "Sometimes (2)", "Usually (3)", and "Always (4)". The total score ranges from 0 to 48. It covers three areas: mouth opening (questions 1, 3, 4, 5, 6), dry mouth (questions 2, 7, 8, 9, 10), and aesthetic concerns (questions 11, 12). Higher scores reflect greater limitations in oral functions.
Fonseca Anamnestic Questionnaire | Two weeks
  Participants are asked to answer 10 questions without any time constraints. Each answer is scored as "yes = 10," "no = 0," and "sometimes = 5." Based on the total score, participants are classified as TMR-Absent (0-15), Mild-TMR (20-40), Moderate-TMR (45-65), and Severe-TMR (70-100).
Modified Hand Mobility in Scleroderma Test (mHAMIS) | Two weeks
  It is a functional test developed specifically for scleroderma to assess an individual's hand function. It evaluates four specific hand movements (finger flexion, finger extension, finger abduction, and dorsal extension). Scores range from 0 (normal) to 3 (complete failure) for each movement, with a total score ranging from 0 to 12.
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Patient | Two weeks
  It is a patient/parent-centered measurement method that helps assess the patient's biopsychosocial aspects, such as disease activity, posture, functional and psychosocial status, fatigue, and school performance. The results from the questions are used to assess the functional status of children, while their psychosocial status is recorded based on their answers to 21 questions (ranging from 0 to 358). A high score indicates a poor psychosocial status.
Juvenile Arthritis Quality of Life Questionnaire (JAQQ) | Two weeks
  It consists of 74 items covering various health domains, including physical functioning, emotional well-being, and general symptoms. The items are divided into four dimensions related to the child's quality of life: gross motor function (GMF), fine motor function (FMF), psychosocial function (PF), and systemic or general symptoms (SGS). Each domain is scored on a Likert-type scale from 1 to 7; higher scores indicate poorer health-related quality of life. There is also a "not applicable to me" option for the items. The scale also includes a pain measurement (10 cm Visual Analog Scale (VAS)) to assess pain, but this score is not included in the total score.
Childhood Health Assessment Questionnaire (CHAQ) | Two weeks
  It assesses the functional abilities of children diagnosed with rheumatic diseases in their daily living activities. It consists of eight subscales (dressing and personal care, standing up, eating, walking, body care, reaching, grasping, activities) (0-3) and also assesses pain and general well-being using a visual analog scale (0-100). A high score indicates low functionality.
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Family | Two weeks
  JAB-Q is a multidimensional questionnaire and a parent (family) form. Developed in Turkish by Ünal and colleagues, the questionnaire is completed by one of the child's parents. The family form evaluates the parents' biopsychosocial status from their own perspective and provides scores ranging from 0 to 102. Higher scores indicate a worse biopsychosocial status.
Pain Catastrophizing Scale-Parent (PCS-P) | Two weeks
  It is assessed using a 5-point Likert scale ranging from 0 (never) to 4 (always) and consists of 13 items. Similar to the child questionnaire, it assesses 3 domains: rumination, magnification, and helplessness. A total score between 0 and 52 is obtained; higher scores reflect a higher level of catastrophizing in parents.
Child and Adolescent Scale of Participation (CASP) | Two weeks
  It is a 20-question survey that evaluates the community participation of children and adolescents in school, neighborhood, and local settings. The survey is divided into four sections: 6 questions about home participation, four questions on neighborhood and community involvement, five questions regarding school participation, and five questions on home and community engagement. It is rated on a scale of "expected for their age (full participation), somewhat limited, very limited, unable to participate, and inapplicable." The survey is completed by the child's family or primary caregiver. The person filling out the questionnaire is asked to select the answer that best describes the child's level of participation. The assessment is scored out of 100 points, with higher scores reflecting a greater level of participation.
Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) | Two weeks
  It was standardized as a biopsychosocial assessment tool and is scored using a 5-point Likert scale, with each item rated from 0 to 4 points. A high total score on the 30-item scale indicates a high level of biopsychosocial impact.
Short Form-36 (SF-36) | Two weeks
  It will be used to determine an individual's quality of life levels. Each sub-parameter is scored between 0 and 100 points, with a high score indicating good health status. The SF-36 scale has eight sub-parameters: general health perception, physical function, social function, pain, mental health, role difficulty due to physical reasons, role difficulty due to emotional reasons, and vitality. It contains 11 questions consisting of a total of 36 items.
Scleroderma Health Assessment Questionnaire (SHAQ) | Two weeks
  It was developed by adding five questions to the HAQ regarding Raynaud's phenomenon, digital ulcers, gastrointestinal, pulmonary, and general scleroderma symptoms, to be rated on a 15 cm line. The SHAQ total score ranges from 0 to 3. A high score indicates low functionality.
Central Sensitization Scale (CSS) | Two weeks
  It is a 40-item scale, scored on a 0-4 Likert scale, that assesses symptoms related to central sensitization. A score above 40 is interpreted as an indicator of central sensitization.
Hospital Anxiety and Depression Scale (HADS) | Two weeks
  It consists of fourteen questions, with odd-numbered questions assessing anxiety and even-numbered questions assessing depression. The options are scored from 0 to 3, with higher scores indicating a worse emotional state. The Turkish cut-off values for the scale are 10 for the anxiety subscale and 7 for the depression subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No